CLINICAL TRIAL: NCT00115284
Title: An Evaluation of Changes in Physician Performance Through Continuous Professional Development
Brief Title: Changes in Physician Performance Through Continuous Professional Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: F10011
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Asthma; Health Personnel
Keywords: Asthma; Education, Medical, Continuing; American Board of Internal Medicine; Recertification; Continuous Professional Development; Practice improvement
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Behavioral: ABIM asthma practice improvement module

SUMMARY:
The purpose of this study is to determine whether having physicians evaluate their management of certain diseases as part of board recertification results in improved patient care.

DETAILED DESCRIPTION:
In the year 2000, the American Board of Internal Medicine introduced continuous professional development as part of its board recertification process. The purpose of these changes were to achieve the following goals:

* To improve the quality of patient care;
* To affirm the high standards expected of a self-regulating, accountable profession;
* To foster continuing scholarship and self-improvement;
* To offer diplomats a portfolio of credentials attesting to competence; and
* To add value to the health care system.

The most notable change in the new recertification process was the addition of practice improvement modules (PIMs). These modules require physicians to review how well they manage a particular chronic disease within their practice and to develop an improvement plan for their practice. In April 2005, it became a requirement that all internists complete a PIM as part of board recertification.

Currently, it not known whether having physicians evaluate their management of certain diseases as part of board recertification will achieve its intended goal of improving patient care. Therefore, the purpose of this trial is to assess whether practice improvement modules result in improved clinical performance.

The PIM selected for this study will focus on asthma. As PIMs seek to improve the quality of care within a practice, the unit of randomization in this study will be clinics (i.e., practices) within the Henry Ford Health System. We will enroll practicing, board-certified internists within the Henry Ford Medical Group (~40 internists or 20 per arm). Clinics (~16 or 8 per arm) will then be randomized to either complete the PIM or not complete the PIM. Participating internists at a site randomized to complete the PIM will be encouraged to work together to complete the asthma PIM. Participating internists at control sites will continue usual care and will not be asked to complete an asthma PIM.

Comparisons: We will assess differences in asthma care by prospectively surveying patients seen by physicians in the intervention group and control group following the intervention period. These analyses will be adjusted by the baseline characteristics of asthma patients seen by participating physicians.

ELIGIBILITY:
Inclusion Criteria:

* Previously board-certified in internal medicine
* Practicing general internist within the Henry Ford Medical Group

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-01; Primary Completion 2006-07 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
1) The proportion of patients prescribed inhaled corticosteroids

SECONDARY OUTCOMES:
1) The proportion of patients reporting instruction on the proper inhaler technique
2) The proportion of patients reporting that asthma triggers were discussed
3) The proportion of patients instructed to use short-acting beta-agonists as needed.
4) The proportion of patients instructed to use a peak flow meter
5) The proportion of patients who received a written action plan for exacerbations
6) The proportion of patients reporting nocturnal asthma symptoms in the past month
7) The proportion of patients reporting regular use of a rescue inhaler daily.

CONTACTS AND LOCATIONS:
Overall Officials: L. Keoki Williams, MD, MPH, Principal Investigator — Center for Health Services Research, Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Benson JA Jr. Certification and recertification: one approach to professional accountability. Ann Intern Med. 1991 Feb 1;114(3):238-42. doi: 10.7326/0003-4819-114-3-238. PMID 1984748
- [Background] Glassock RJ, Benson JA Jr, Copeland RB, Godwin HA Jr, Johanson WG Jr, Point W, Popp RL, Scherr L, Stein JH, Taunton OD. Time-limited certification and recertification: the program of the American Board of Internal Medicine. The Task Force on Recertification. Ann Intern Med. 1991 Jan 1;114(1):59-62. doi: 10.7326/0003-4819-114-1-59. No abstract available. PMID 1983934
- [Background] Wasserman SI, Kimball HR, Duffy FD. Recertification in internal medicine: a program of continuous professional development. Task Force on Recertification. Ann Intern Med. 2000 Aug 1;133(3):202-8. doi: 10.7326/0003-4819-133-3-200008010-00012. PMID 10906835
- [Background] Norcini JJ, Lipner R, Downing SM. How meaningful are scores on a take-home recertification examination? Acad Med. 1996 Oct;71(10 Suppl):S71-3. doi: 10.1097/00001888-199610000-00048. No abstract available. PMID 8940939
- [Background] Norcini JJ, Lipner RS. Recertification: is there a link between take-home and proctored examinations? Acad Med. 1999 Oct;74(10 Suppl):S28-30. doi: 10.1097/00001888-199910000-00031. No abstract available. PMID 10536585
- [Background] Kassirer JP. ABIM looks toward the future. Am J Med. 1996 Feb;100(2):123-4. doi: 10.1016/s0002-9343(97)89448-x. No abstract available. PMID 8629644
- [Background] Campbell C, Parboosingh J, Gondocz T, Babitskaya G, Pham B. A study of the factors that influence physicians' commitments to change their practices using learning diaries. Acad Med. 1999 Oct;74(10 Suppl):S34-6. doi: 10.1097/00001888-199910000-00033. No abstract available. PMID 10536587
- [Background] Davis DA, Thomson MA, Oxman AD, Haynes RB. Changing physician performance. A systematic review of the effect of continuing medical education strategies. JAMA. 1995 Sep 6;274(9):700-5. doi: 10.1001/jama.274.9.700. PMID 7650822
- [Derived] Simpkins J, Divine G, Wang M, Holmboe E, Pladevall M, Williams LK. Improving asthma care through recertification: a cluster randomized trial. Arch Intern Med. 2007 Nov 12;167(20):2240-8. doi: 10.1001/archinte.167.20.2240. PMID 17998498